CLINICAL TRIAL: NCT06599931
Title: CEREBELLO-MOTOR NEUROMODULATION AFTER STROKE
Brief Title: Cerebello-motor Neuromodulation After Stroke. CERSTIM.
Acronym: CERSTIM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: C23-100; 2024-A00623-44 (Registry Identifier: IDRCB)
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Stroke; Healthy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Three sessions active tACS 20 minutes, 50Htz active tACS 20 minutes, 70 Htz sham
  Order will be randomized
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are blinded from the type of intervention (sham, 50 Htz or 70 Htz)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- tACS session 50 Hz (Active Comparator): Three single sessions of tACS, each lasting 20 minutes, will be conducted 7-15 days apart, with a different frequency (50 or 70 Hz, corresponding to gamma oscillations) or a placebo frequency known as "sham."
  Interventions: Device: tACS Transcranial alternating stimulation
- tACS session 70 Hz (Active Comparator): Three single sessions of tACS, each lasting 20 minutes, will be conducted 7-15 days apart, with a different frequency (50 or 70 Hz, corresponding to gamma oscillations) or a placebo frequency known as "sham."
  Interventions: Device: tACS Transcranial alternating stimulation
- tACS Sham session (Sham Comparator): Three single sessions of tACS, each lasting 20 minutes, will be conducted 7-15 days apart, with a different frequency (50 or 70 Hz, corresponding to gamma oscillations) or a placebo frequency known as "sham."
  Interventions: Device: tACS Transcranial alternating stimulation

INTERVENTIONS:
Device: tACS Transcranial alternating stimulation — session of 20 minutes

SUMMARY:
The CERSTIM study is a physiopatholgical study investigating transcranial alternating current stimulation in stroke patients in the cerebello-motor loop.

The design is a cross over design testing two frequencies in the gamma band and one placebo.

We will use behavioural data, functional MRI, and Electroencephalography to disentangle the effect of tACS and its frequency.

Healthy participants will be also recruited.

DETAILED DESCRIPTION:
Neuromodulation, by the means of Non-Invasive Brain Stimulation techniques, is a promising method to enhance motor recovery of the upper limb following a stroke. However, none of these techniques have yet been effectively transferred to the patient's bedside. An international group of experts has examined this issue, identifying barriers that need to be overcome for successful transferability. Among their findings, two were particularly emphasized: (i) the insufficient characterization of the mechanisms through which these stimulations are effective, and (ii) the comparison of stimulation parameters before moving on to larger samples. We have decided to use this model to study tACS (transcranial Alternating Current Stimulation) on the cerebellomotor network.

The choice of tACS is justified by (i) its ability to "entrain" a neural network through its oscillations, (ii) its innovative nature, and (iii) its "wearable" characteristic, making it quickly transferable. The choice of the cerebellomotor network is based on literature data showing that (i) the cerebellum plays a crucial role in motor learning in healthy individuals (which is one of the substrates of post-stroke recovery), and (ii) cerebellomotor synchronization is a good prognostic indicator for the recovery of hand motor function.

In light of these findings, we have decided to conduct a pathophysiological, bi-centric study to determine the cerebral mechanisms by which tACS acts on the cerebellomotor network. Three single sessions of tACS, each lasting 20 minutes, will be conducted 7-15 days apart, with a different frequency (50 or 70 Hz, corresponding to gamma oscillations) or a placebo frequency known as "sham." To understand the cerebral mechanisms, we will use Magnetic Resonance Imaging (MRI) and Electroencephalography (EEG). We will also examine a behavioral motor adaptation task on a tablet. The order in which the three frequencies are applied will be randomized This study will include 30 patients and 15 healthy subjects. The patients will be individuals who have suffered a stroke more than 6 months ago, resulting in a hand deficit without complete paralysis. The healthy controls will serve as a reference for mechanisms and imaging/electrophysiology data.

We hypothesize the following: The mechanisms involved following cerebellomotor stimulation could include a modification of brain rhythms in the beta or gamma band during movement, an increase in activity in the primary motor cortex, or a change in the excitation-inhibition balance between the cerebellum and the primary motor cortex, or directly at the level of the primary motor cortex. These different mechanisms may vary depending on the frequency used.

This research is part of the NEUROTECH Impulse Program managed by INSERM.

ELIGIBILITY:
PATIENTS

Inclusion Criteria:

* Male or female aged 18 years or older on the day of inclusion.
* Affiliated with a social security system, Universal Health Coverage (CMU), or any equivalent scheme.
* Ischemic stroke or intraparenchymal hematoma that occurred more than 6 months ago, with no upper time limit.
* Motor deficit of the upper limb confirmed by the ARAT scale, with the ability to grip and press on a tablet.
* stroke lesion not affecting the motor cortex in the hand knob area.

Exclusion Criteria:

-- Pregnant and breastfeeding women

* Total paralysis of the affected hand
* Conditions that are life-threatening or could compromise follow-up during the study period
* Contraindications to MRI and tACS (ferromagnetic surgical clips, ocular implants, intraocular or nervous system metallic foreign bodies, implants or metallic objects likely to concentrate the radiofrequency field, cochlear implants, brain or cardiac stimulators, presence of a craniotomy scar)
* Participation in another biomedical study focused on motor or overall recovery during the same period, or current exclusion period from another biomedical study

HEALTHY

Inclusion Criteria:

* Male or female aged 18 years or older on the day of inclusion.
* Affiliated with a social security system, Universal Health Coverage (CMU), or any equivalent scheme.

Non inclusion criteria

-- Pregnant and breastfeeding women

* Conditions that are life-threatening or could compromise follow-up during the study period
* Contraindications to MRI and tACS (ferromagnetic surgical clips, ocular implants, intraocular or nervous system metallic foreign bodies, implants or metallic objects likely to concentrate the radiofrequency field, cochlear implants, brain or cardiac stimulators, presence of a craniotomy scar)
* Participation in another biomedical study during the same period, or current exclusion period from another biomedical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-12-13 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
change in activation in the primary motor cortex and cerebellum using functional magnetic Resonance | [Time Frame: within 1 hour before and after the intervention]
  The activity of cerebellomotor regions is measured in functional task MRI with a hand motor task performed in the machine (squeezing a handle).
  The average BOLD signal in the cerebellum and M1 regions is measured using a general linear model adapted to functional MRI images such as SPM and its toolboxes.

SECONDARY OUTCOMES:
comparison between activation in the primary motor cortex and cerebellum using functional magnetic Resonance with the 50 Htz versus the 70 Htz frequency | [Time Frame: within 1 hour before and after the intervention]
  The measurement method is identical to that used for the primary endpoint. Only the final statistical test changes (comparison of differences between each session).
  final change statistics (comparison of difference between each session).
change in functional connectivity between the primary motor cortex and cerebellum using functional magnetic Resonance | [Time Frame: within 1 hour before and after the intervention]
  The measurement method is based on functional task MRI. It involves a z-score of the correlation between the signal of 2 regions in time belonging to the motor network.
change in functional connectivity using EEG after intervention and comparison between frequencies of tACS | [Time Frame: within 1 hour before and after the intervention]
  The measurement method will be functional connectivity measured by an index called wSMI (weighted-Symbolic Mutual Information), which is an EEG marker. EEG data will be collected via the Starstim Neuroelectrics system and analyzed using in-house scripts (developed in-house) in Matlab and Python before and after each session, and we will also compare differences in change between the two sessions.
change in behaviour after intervention and comparison between frequencies of tACS | [Time Frame: within 1 hour before and after the intervention]
  behaviour will be assessed on a motor learning task (accuracy, reaction time). The measurement method will be a SRT (serial reaction time) task with visuomotor adaptation where the subject must obey these instructions. Error rate and reaction time will be measured.
  will be measured.
comparison of the prespecified patients outcome with those of healthy subjects | [Time Frame: within 1 hour before and after the intervention]
  All the above measurements will be carried out in a cohort of healthy subjects and compared with patients.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte ROSSO, MD PHD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (2):
- France (2):
  - ICM_ Institut du Cerveau et de la Moelle épinière, Hôpital Pitié, 47 Bd de l'Hôpital, Paris
  - ToNIC - Toulouse neuro Imaging center (Inserm)Pavillon Baudot, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided
IPD could be shared upon request and if RGPD rules are respected and if ethics comittee agrees